CLINICAL TRIAL: NCT02722707
Title: Clinical Use of a Magnetic Anal Sphincter Augmentation Device, Trade Name FENIX. A Humanitarian Use Device ( HUD), Which Has Recently Received a Humanitarian Device Exemption (HDE) From the Food and Drug Administration ( FDA)
Brief Title: Clinical Use of a Magnetic Anal Sphincter Augmentation Device, Trade Name FENIX
Status: No longer available | Type: Expanded Access
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Paul D Pettit, Consultant Gyn Surgery, Mayo Clinic
Other Study IDs: 16-000150
Record Dates: First submitted 2016-02-26; First posted 2016-03-30 (Estimated); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

INTERVENTIONS:
Device: magnetic anal sphincter augmentation for fecal incontinence — Surgical placement of HUD called FENIX for female patients that have failed conservative therapy and less invasive therapies or who are not candidates for such therapies
  Other Names: FENIX

SUMMARY:
This registration is for clinical use of the FENIX, a Humanitarian Use Device (HUD) for fecal incontinence. This device is indicated for the treatment of fecal incontinence in patients who are not candidates for or have previously failed conservative treatment and less invasive therapy options (e.g. bulking agents, radiofrequency ablation, sacral nerve stimulation).

DETAILED DESCRIPTION:
The FENIX is surgically placed. This surgery could be an outpatient procedure or at most an overnight stay in the hospital. The design of the device allows it to be effective immediately. The device is similar to the LINX device used for esophageal reflux. It is a circular set of magnets which surrounds the ano-rectal support. The size of the device is determined at the time of surgery so that the ano-rectum is closed. When the patient strains at stool, this pressure separates the magnets and allows passage of stool. The magnets are held together by an independent malleable titanium wire. Once straining at stool stops, the magnets are able to re-connect or close the rectum. We will monitor patients for postoperative complications related to surgery.

ELIGIBILITY:
Inclusion Criteria:

* non-pregnant female patients
* 18 years of age or older with fecal incontinence
* failed conservative therapy ( pelvic floor physical therapy, medications) and failed trial of interstim.

Exclusion Criteria:

* patients less than 18 years of age,
* pregnant
* previous radiation to pelvis,
* chronic diarrhea or inflammatory bowel disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Paul D Pettit, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota